CLINICAL TRIAL: NCT05572450
Title: An Exploratory Study to Establish the Dose, Safety and Pathogenicity of a New Influenza H1N1 Challenge Strain in Healthy Participants 18 to 55 Years of Age
Brief Title: Dose, Safety, and Pathogenicity of a New Influenza H1N1 Challenge Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvivo (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HRD-vCS-001
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Influenza A H1N1
Keywords: Influenza; Human Challenge Trial; H1N1; Flu
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Infectious Titre 1 (Experimental): Dose Arm 1 (Part A): Approximately 10^5.5 TCID50/mL (titre may be adjusted based on stock titre)
  Interventions: Other: Infectious Titre 1
- Infectious Titre 2 (Experimental): Dose Arm 2 (Part A): Approximately 10^4.5 TCID50/mL (titre may be adjusted based on stock titre)
  Interventions: Other: Infectious Titre 2
- Infectious Titre 3 (Experimental): Optional Dose Arm 3 (Part B): to be determined (TBD), depending on outcome of Part A
  Interventions: Other: Infectious Titre 3
- Infectious Titre 4 (Experimental): Optional Dose Arm 4 (Part B): TBD, depending on outcome of Part A
  Interventions: Other: Infectious Titre 4

INTERVENTIONS:
Other: Infectious Titre 1 — Approximately 10^5.5 TCID50/mL (titre may be adjusted based on stock titre)
  Arms: Infectious Titre 1
Other: Infectious Titre 2 — Approximately 10^4.5 TCID50/mL (titre may be adjusted based on stock titre)
  Arms: Infectious Titre 2
Other: Infectious Titre 3 — To be determined (TBD), depending on outcome of Part A
  Arms: Infectious Titre 3
Other: Infectious Titre 4 — TBD, depending on outcome of Part A
  Arms: Infectious Titre 4

SUMMARY:
A total of up to 90 participants may be given H1N1 influenza challenge virus.

In Part A, 40 participants will be randomly allocated to one of two groups to be given one of two virus doses (Virus Dose 1 or Virus Dose 2).

Based on the outcome of Part A, participants in Part B, may be given Virus Dose 1, Virus Dose 2, or another virus dose (e.g., Virus Dose 3)

DETAILED DESCRIPTION:
Influenza viruses are associated with significant human disease and cause annual epidemics during autumn and winter. Although most people recover within 1 to 2 weeks without requiring medical attention, seasonal influenza yearly results in approximately 3 to 5 million cases of severe illness and up to 500,000 deaths worldwide, particularly among the very young, elderly, and chronically ill.

The H1N1 virus used for the challenge virus originated from a cell-culture derived candidate vaccine virus (ccCVV), provided by the Centers for Disease Control an Prevention (CDC) in the USA.

In Part A, 40 participants will be randomly allocated to one of two groups to be given one of two virus doses (Virus Dose 1 or Virus Dose 2).

Based on the outcome of Part A, participants in Part B, may be given Virus Dose 1, Virus Dose 2, or another virus dose (e.g., Virus Dose 3)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult male or female aged between 18 and 55 years
* A total body weight ≥50 kg and body mass index (BMI) ≥18 kg/m2 and ≤35kg/m2
* In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety.
* Documented medical history
* Adherence to contraception requirements
* Serosuitable for the challenge virus.

Exclusion Criteria:

* History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract (LRT) infection within 4 weeks prior to the first study visit.
* Any history or evidence of any clinically significant or currently active disease.
* Any participants who have smoked ≥10 pack years at any time.
* Female participants who are breastfeeding, or have been pregnant within 6 months prior to the study, or have a positive pregnancy test at any point during screening or prior to inoculation.
* Lifetime history of anaphylaxis and/or a lifetime history of severe allergic reaction.
* Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
* Significant abnormality of the nose, epistaxis, nasal or sinus surgery.
* Recent vaccinations or intention to receive vaccination before the final follow up visit.
* Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned inoculation or planned during the 3 months after the final visit.
* Recent receipt of investigational drugs or challenge viruses.
* Use or anticipated use during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows.
* Positive drugs of abuse test or recent history or presence of alcohol addiction
* A forced expiratory volume in 1 second (FEV1) <80%.
* Positive HIV, hepatitis B virus, or hepatitis C virus test.
* Presence of fever, defined as participant presenting with a temperature reading of ≥37.9C on Day -2/-1 and/or pre-inoculation on Day 0.
* Those employed or immediate relatives of those employed at hVIVO or the sponsor.
* Any other reason, in the opinion of the investigator deems the participant unsuitable for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
To determine the safe and optimal titre of the influenza challenge virus | Day 0 to Day 28
  To identify a safe and infectious dose of wild-type influenza virus in healthy participants, suitable for future intervention studies that:
  • Has an acceptable safety profile as measured by:
  Occurrence of adverse events (AEs) related to the viral challenge
  Occurrence of serious AEs (SAEs) related to the viral challenge
  Induces laboratory-confirmed infection in ≥40% of inoculated participants (ideally between 50% and 80%).

CONTACTS AND LOCATIONS:
Overall Officials: Alex Mann, Study Director — hVIVO Services Ltd.
Locations (1):
- hVIVO Services Ltd, London, United Kingdom